CLINICAL TRIAL: NCT05450874
Title: A Novel MSE Score to Predict the Postoperative Prognosis of Patients With Ruptured Hepatocellular Carcinoma
Brief Title: A Novel MSE Score to Predict rHCC Patients
Status: Completed | Type: Observational
Sponsor: Tongji Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2019CFB433
Record Dates: First submitted 2022-07-05; First posted 2022-07-11 (Actual); Last update posted 2022-07-11 (Actual); Status verified 2022-06

CONDITIONS: HCC
MeSH Terms: interventions — Hepatectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Training cohort
  Interventions: Procedure: hepatectomy
- Validation cohort
  Interventions: Procedure: hepatectomy

INTERVENTIONS:
Procedure: hepatectomy

SUMMARY:
Develop and validate a novel scoring system based on pathological factors to predict the postoperative survival of patients with rHCC.Patients with rHCC who underwent hepatectomy were recruited from two hospitals.Exploring whether this scoring system is related to prognosis

ELIGIBILITY:
Inclusion Criteria:

* a diagnosis of ruptured tumor confirmed by enhanced computed tomography (CT) and/or abdominal magnetic resonance imaging (MRI),
* a diagnosis of HCC made by two experienced pathologists

Exclusion Criteria:

* extrahepatic HCC metastasis
* death within 1 month after surgery

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 221 patients with rHCC who underwent liver resection from February 2010 to March 2016 at Tongji Hospital and 97 patients with rHCC who underwent hepatectomy at Zhongshan People's Hospital during the same period were included in this study
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2010-02-01 (Actual); Primary Completion 2017-03-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
overall survival | 2010-2022
  Time from the first postoperative day to survival at the last follow-up

IPD SHARING:
Plan to Share IPD: Undecided